CLINICAL TRIAL: NCT03834987
Title: NGLY1 Deficiency: A Prospective Natural History Study
Status: Terminated | Type: Observational
Why Stopped: Study concluded by Stanford University
Sponsor: Stanford University (Other)
Collaborators: Grace Science Foundation (Other)
Responsible Party: Principal Investigator, Maura Ruzhnikov, Clinical Assistant Professor, Stanford University
Other Study IDs: IRB-47335
Record Dates: First submitted 2019-01-23; First posted 2019-02-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Genetic Syndrome
Keywords: NGLY1 Deficiency
MeSH Terms: conditions — Genetic Diseases, Inborn; NGLY1 deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine and blood samples.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Neurodevelopmental Assessment — Developmental assessment at baseline and longitudinally as measured by age and ability-appropriate scales, including: the Mullen Scales of Early Learning, the Peabody Scales of Motor Development, the Vineland 3, and Beery Visual Motor Integration

SUMMARY:
NGLY1 deficiency is a rare genetic disorder that is characterized by: global developmental delay and/or intellectual disability, hypo- or alacrima, transient elevation of transaminases, and a hyperkinetic movement disorder. Significant phenotypic variability has been observed in the small number of affected individuals described in the medical literature.

The purpose of this study is to describe the natural history of NGLY1 deficiency in a prospective, detailed, and highly uniform manner. Study participants will be closely monitored over the course of five years in order to:

* understand the clinical spectrum and progression of NGLY1 deficiency using standardized clinical and neurodevelopmental assessments
* identify clinical and biomarker endpoints for use in therapeutic trials, and
* identify genotype-phenotype correlations

Close clinical follow-up will allow for generation of a rich dataset and detailed understanding of the natural history of NGLY1 deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Parent(s)/legal representative and/or participant must be willing and able to give informed consent/assent for participation in the study
* Males or females of any age
* Suspected or confirmed diagnosis of NGLY1 deficiency with genetic variants in both NGLY1 alleles and consistent clinical characteristics
* Participant and caregiver must be willing to provide clinical data, participate in standardized assessments, and provide biological samples (if living in the United States)
* Willingness to travel to Palo Alto, CA is favored, but not required

Exclusion Criteria:

* The presence of a second, confirmed disorder, genetic or otherwise, affecting neurodevelopment or with other overlapping symptoms of NGLY1 deficiency

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals of any age with NGLY1 deficiency.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-11-19 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Detailed phenotyping of the clinical course of NGLY1 deficiency over time | 5 years
  Conducted in patients with NGLY1 deficiency: detailed standardized general, neurologic, dysmorphologic, and ophthalmologic evaluations; clinical laboratory studies; electroencephalogram; nerve conduction studies; quantitative studies of autonomic function; scoring of movement disorder and NGLY1 deficiency symptom scales; and a timed 10-meter walk test. As much information as available will also be collected from existing medical records including clinical evaluations, imaging studies and neuropsychological and motor function evaluations.
Neurodevelopmental profile of NGLY1 deficiency as measured using Mullen Scales of Early Learning | 5 years
  Developmental assessment at baseline and longitudinally, if age and ability-appropriate.
Neurodevelopmental profile of NGLY1 deficiency as measured using Bruininks-Oseretsky Test of Motor Proficiency, Second Edition | 5 years
  Developmental assessment at baseline and longitudinally, if age and ability-appropriate.
Neurodevelopmental profile of NGLY1 deficiency as measured using the Peabody Scales of Motor Development | 5 years
  Developmental assessment at baseline and longitudinally, if age and ability-appropriate.
Neurodevelopmental profile of NGLY1 deficiency as measured using the Differential Ability Scales II | 5 years
  Developmental assessment at baseline and longitudinally, if age and ability-appropriate.
Neurodevelopmental profile of NGLY1 deficiency as measured using the Beery Visual Motor Integration developmental test | 5 years
  Developmental assessment at baseline and longitudinally, if age and ability-appropriate.

SECONDARY OUTCOMES:
Participant quality of life as measured through the Pediatric Quality of Life Inventory (PedsQL) | 5 years
  Quality of life will be evaluated at baseline and longitudinally.
Caregiver quality of life as measured through the 36 Item Short Form Survey (SF36) | 5 years
  Quality of life will be evaluated at baseline and longitudinally. Caregivers will complete the survey but will not be enrolled in the study.
Biomarkers for NGLY1 deficiency identified during the course of the study | 5 years
  Longitudinal collection and monitoring of laboratory studies and clinical presentation as measured through standardized and quantitative assessments may identify biomarkers for NGLY1 deficiency.

CONTACTS AND LOCATIONS:
Overall Officials: Maura Ruzhnikov, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers and clinicians with academic interest in NGLY1 deficiency may be provided access to data obtained through this study. Any data or samples shared outside of Stanford University will be done so in a coded fashion with no protected health information included and with the execution of all applicable agreements (i.e. a material transfer agreement) or ongoing collaborations as approved in eProtocol 47335.

REFERENCES:
- [Result] Levy RJ, Frater CH, Gallentine WB, Phillips JM, Ruzhnikov MR. Delineating the epilepsy phenotype of NGLY1 deficiency. J Inherit Metab Dis. 2022 May;45(3):571-583. doi: 10.1002/jimd.12494. Epub 2022 Mar 11. PMID 35243670
- [Derived] Frater CH, Ruzhnikov MRZ, Beres S, Alcorn D, Shue A, Levy RJ. Ocular features of NGLY1 deficiency from a prospective longitudinal cohort. J AAPOS. 2024 Jun;28(3):103925. doi: 10.1016/j.jaapos.2024.103925. Epub 2024 Apr 30. PMID 38697387
- See also: Grace Science Foundation — https://gracescience.org/
- See also: Neurogenomics at Stanford — https://www.stanfordchildrens.org/en/service/neurogenomics